CLINICAL TRIAL: NCT05004077
Title: Repeated Amiodarone Dosing In Cardiac surgicaL Procedures
Acronym: RADICAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: limited enrollment
Sponsor: Kevin W Hatton, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Kevin W Hatton, MD, PhD, Professor, Dept of Anesthesiology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67919
Record Dates: First submitted 2021-08-02; First posted 2021-08-13 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Conventional amiodarone dosing regimen (CDR) (Active Comparator): Initial amiodarone bolus of 150 mg IV over 10 minutes then a 24-hour amiodarone loading infusion (1 mg/min for 6 hours followed by 0.5 mg/min for 18 hours), followed by enteral (400 mg amiodarone oral or per tube three times daily or 2 times daily if the patient has gastrointestinal intolerance when taking the drug three times daily) or intravenous amiodarone (0.5 mg/min continuous infusion) to complete an 8-gm total amiodarone load. Maintenance amiodarone (200 mg amiodarone oral or per tube once daily) at discretion of attending physician.
  Interventions: Drug: AMIODARONE
- Repeated amiodarone bolus dosing regimen (RBDR) (Active Comparator): Initial amiodarone bolus of 150 mg IV over 10 minutes, then 1.0 mg/min IV amiodarone infusion for 6 hours, then a 0.5 mg/min IV amiodarone infusion for 18 hours, followed by enteral (400 mg amiodarone oral or per tube three times daily or 2 times daily if the patient has gastrointestinal intolerance when taking the drug three times daily) or intravenous amiodarone (0.5 mg/min continuous infusion) to complete an 8-gm total amiodarone load. In addition, patients in the RBDR will receive an additional 150 mg IV amiodarone bolus whenever the patient develops tachycardia (Heart Rate (HR) = 110 beats per minute) lasting more than 10 minutes. This bolus may be repeated up to a total of 5 times (6 total boluses) over the first 24 hours. Maintenance amiodarone (200 mg amiodarone oral or per tube once daily) at discretion of attending physician.
  Interventions: Drug: AMIODARONE

INTERVENTIONS:
Drug: AMIODARONE — Assess the effectiveness of different dosing strategies of amiodarone.

SUMMARY:
This study is a single-center, prospective, randomized, open-label trial of subjects who develop atrial fibrillation after non-emergent cardiac surgery at the University of Kentucky Chandler Medical Center (UKCMC). Patients will be randomized to receive either a conventional amiodarone dosing regimen (CDR) or a repeated amiodarone bolus dosing regimen (RBDR).

DETAILED DESCRIPTION:
This study will screen and consent approximately 150 patients undergoing non-emergent cardiac surgery. Approximately 60 of these patients are likely to develop stable postoperative atrial fibrillation (POAF) in the postoperative period. Amiodarone is commonly given as an initial intravenous (IV) bolus (150 mg IV) followed by a combined IV and oral load to a total dose of 8 gm. Because of amiodarone's beta-blocker activity, the IV bolus in patients with POAF is associated with a reduced heart rate that may lead to restoration of NSR. For this reason, some clinicians will provide up to 5 additional IV amiodarone boluses during the drug's loading period to treat RVR.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years old or older
* Subject must be willing to give written informed consent
* Subject must undergo or scheduled for non-emergent cardiac surgery, including coronary artery bypass grafting (CABG), non-infectious valve repair or replacement, atrial or septal defect repair, thoracic aortic replacement surgery, or any combination of these procedures

Exclusion Criteria:

* Documented allergy to amiodarone or iodine
* History of atrial fibrillation or other heart conduction system abnormality
* History of cardiac maze, pulmonary vein isolation, or other procedure affecting the conduction system
* Scheduled cardiac maze, pulmonary vein isolation, or other procedure affecting the conduction system
* Low cardiac index or cardiogenic shock requiring pharmacologic or mechanical support
* History of pre-existing respiratory system disease requiring oxygen therapy prior to admission
* History of cirrhosis or other chronic liver diseases
* Pregnancy or breastfeeding mothers
* Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hatton, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR) | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Normal Sinus Rhythm -24 HRS
Description: Percentage of patients who develop stable POAF after non-emergent cardiac surgery, the percentage of patients who have converted to NSR at 24-hours after receiving a repeated amiodarone bolus and loading dose regimen to the percentage of patients who have converted to NSR after a conventional amiodarone IV loading dose regimen.
Time Frame: 24-hours after receiving amiodarone bolus
Population: No data released because enrollment was three participants, and one group had a singular participant. Therefore, confidentiality of the participant's health information could be impacted if the outcome measures were displayed.for that group with only one participant. Additionally, the other group only had two participants, again, release of this information could impact their right to confidentiality.
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Total Target Heart Rate Time
Description: Total time, in minutes, during the first 24 hours that the patient achieves target HR (HR < 110 bpm) between patients who receive a repeated amiodarone bolus dosing regimen and those who receive a conventional amiodarone bolus dosing regimen
Time Frame: 24-hours after receiving amiodarone bolus
Population: as for outcome 1
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Target Heart Rate
Description: Time to achieve target HR (HR < 110 bpm) between patients who receive a repeated amiodarone bolus dosing regimen and those who receive a conventional amiodarone bolus dosing regimen
Time Frame: 24-hours after receiving amiodarone bolus
Population: as for outcome 1
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Normal Sinus Rhythm -Hospital Index
Description: Percentage of patients who achieve NSR by ICU discharge and hospital discharge between patients who receive a repeated amiodarone bolus dosing regimen and those who receive a conventional amiodarone bolus dosing regimen
Time Frame: duration of ICU and hospital visit, up to 20 days
Population: as for outcome 1
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Recurrent AF
Description: Percentage of patients who have recurrent AF before ICU discharge and before hospital discharge and patients who receive a repeated amiodarone bolus dosing regimen and those who receive a conventional amiodarone bolus dosing regimen
Time Frame: duration of ICU and hospital visit, up to 20 days
Population: as for outcome 1
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection period is during hospitalization, approximately 5 days.
Arm/Group | Conventional Amiodarone Dosing Regimen (CDR) | Repeated Amiodarone Bolus Dosing Regimen (RBDR)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT05004077/Prot_002.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT05004077/SAP_003.pdf